CLINICAL TRIAL: NCT00469014
Title: Busulfan-Fludarabine-Clofarabine With Allogeneic Stem Cell Transplantation for Advanced Refractory Acute Myeloid Leukemia, Myelodysplastic Syndrome, and Advanced, Gleevec Refractory Chronic Myeloid Leukemia. A Randomized Phase II Study.
Brief Title: Busulfan, Fludarabine, Clofarabine With Allogeneic Stem Cell Transplantation for Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0200
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Myelodysplastic Syndrome; MDS; Chronic Myeloid Leukemia; CML; Busulfan; Busulfex; Myleran; Fludarabine; Fludara; Fludarabine Phosphate; Clofarabine; Clofarex; Clolar; Allogeneic stem cell transplantation; ASCT; Stem Cell; Gleevec; Imatinib Mesylate
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Clofarabine; Busulfan; fludarabine; fludarabine phosphate; Bone Marrow Transplantation; thymoglobulin; Antilymphocyte Serum; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine (Active Comparator): 4-day Treatment Period Day -6 to Day -2: Busulfan 30 mg/m^2 intravenous (IV) Daily + Fludarabine 30 mg/m^2 IV Daily; + Clofarabine 10 mg/m^2 IV Daily; Thymoglobulin Day -3 to Day -1, and Stem Cell Infusion Day 0.
  Interventions: Drug: Clofarabine; Drug: Busulfan; Drug: Fludarabine; Other: Stem Cell Infusion; Drug: Thymoglobulin (ATG); Drug: Filgrastim
- Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine (Experimental): 4-day Treatment Period Day -6 to Day -2: Busulfan 20 mg/m^2 IV + Fludarabine 20 mg/m^2 IV Daily + Clofarabine 20 mg/m^2 IV Daily. Thymoglobulin Day -3 to Day -1, and Stem Cell Infusion Day 0.
  Interventions: Drug: Clofarabine; Drug: Busulfan; Drug: Fludarabine; Other: Stem Cell Infusion; Drug: Thymoglobulin (ATG); Drug: Filgrastim
- Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine (Experimental): 4-day Treatment Period Day -6 to Day -2: Busulfan 10 mg/m^2 IV Daily + Fludarabine 10 mg/m^2 IV Daily + Clofarabine 30 mg/m^2 IV Daily. Thymoglobulin Day -3 to Day -1, and Stem Cell Infusion Day 0.
  Interventions: Drug: Clofarabine; Drug: Busulfan; Drug: Fludarabine; Other: Stem Cell Infusion; Drug: Thymoglobulin (ATG); Drug: Filgrastim
- Arm 4: Busulfan + Clofarabine (Experimental): 4-day Treatment Period Day -6 to Day -2: Busulfan 40 mg/m^2 IV Daily + Clofarabine 40 mg/m^2 IV Daily. Thymoglobulin Day -3 to Day -1, and Stem Cell Infusion Day 0.
  Interventions: Drug: Clofarabine; Drug: Busulfan; Other: Stem Cell Infusion; Drug: Thymoglobulin (ATG); Drug: Filgrastim

INTERVENTIONS:
Drug: Clofarabine — Day -6 to Day -3 for Arm 1 = 10 mg/m^2 intravenous (IV) Daily; Arm 2 = 20 mg/m^2 IV Daily; Arm 3 = 30 mg/m^2 IV Daily; Arm 4 = 40 mg/m^2 IV Daily
  Other Names: Clofarex; Clolar
Drug: Busulfan — Day -6 to Day -3 for Arm 1: 30 mg/m^2 IV Daily; Arm 2: 20 mg/m^2 IV Daily; Arm 3: 10 mg/m^2 IV Daily; Arm 4: 40 mg/m^2 IV Daily.
  Test dose Day -8 32 mg/ m^2 IV over 45 min, rest on Day -7.
  Other Names: Busulfex; Myleran
Drug: Fludarabine — Day -6 to Day -3 for Arm 1: 30 mg/m^2 IV Daily; Arm 2: 20 mg/m^2 IV Daily; Arm 3: 10 mg/m^2 IV Daily
  Other Names: Fludarabine Phosphate; Fludara
  Arms: Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine; Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine; Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine
Other: Stem Cell Infusion — Day 0 stem cell infusion (Bone marrow or peripheral blood progenitor cells (PBPC))
  Other Names: Bone Marrow Transplant; BMT; peripheral blood progenitor cells; PBPC; Unstimulated bone marrow transplant; bone marrow transplantation; ABM transplantations; autologous bone marrow transplantation
Drug: Thymoglobulin (ATG) — Day -3 to Day -1 at 0.5 mg/kg IV on Day -3; 1.5 mg/kg on Day -2 and 2.0 mg/kg on Day -1.
  Other Names: Thymoglobulin; Antithymocyte Globulin
Drug: Filgrastim — Subcutaneous injection daily, starting 1 week after Stem Cell Transplant.
  Other Names: G-CSF; Granulocyte colony-stimulating factor; GCSF

SUMMARY:
The goal of this clinical research study is to find the best dose of clofarabine and fludarabine that can be given with busulfan followed by an allogeneic blood stem cell transplant. Researchers will study whether this combination can help to control the disease, and look at the safety of this combination. Researchers also want to find out if combining busulfan with clofarabine alone or combining busulfan with both fludarabine and clofarabine will improve the treatment, compared with the previous standard method using busulfan and fludarabine alone.

DETAILED DESCRIPTION:
Busulfan is a chemotherapy drug that kills cancer cells by binding to DNA (the genetic material of cells). Clofarabine is designed to interfere with the growth and development of cancer cells. Fludarabine is designed to interfere with DNA repair enzymes so that the leukemic cells cannot repair damaged DNA. This may increase the likelihood of the cell dying. These drugs are being given to try to kill cancerous cells and weaken your immune system in order to lower the risk of stem cell transplant rejection.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 4 study groups. Three (3) of the groups will receive busulfan, fludarabine, and clofarabine at different dose levels. The 4th group will only receive busulfan and clofarabine. As the study continues, participants will be assigned using a method called adaptive randomization. This method works by increasing the chances of being assigned to the group that has had the best results in the study so far. You will know which group you have been assigned to.

Participants will receive busulfan, fludarabine, and/or clofarabine once a day for 4 doses. You will first receive an additional low-level "test" dose of busulfan given by vein to check how your blood levels change over time. This information will be used to decide the next dose needed to reach a target blood level of busulfan. You will have a total of about 6 and 1/2 tablespoons of blood drawn over time to check your busulfan blood levels following one or more of the busulfan treatments. Up to 11 samples of blood will be drawn to check your blood levels of busulfan during the next 11 hours following the test dose and the first high-dose busulfan treatment. Each sample will require about 1 teaspoon of blood. A heparin lock line will be placed in a vein to lower the number of needle sticks needed for these draws. If it is not possible for these blood level tests to be performed for technical or scheduling reasons, you will receive the standard fixed (unchanging) dose of busulfan.

Clofarabine and fludarabine (if applicable) will be given through a central venous catheter (CVC) over 1 hour, once a day, for 4 days. Busulfan will also be given through the CVC over 3 hours.

If you are going to be receiving a transplant from an HLA-nonidentical or unrelated donor, you will also receive thymoglobulin (ATG) over 4 hours on the 3 days before the transplant to further weaken your immune system to reduce the risk of rejecting of the transplant. After the transplant, you will receive tacrolimus, methotrexate, or other immunosuppressive (lowering the immune system) drugs in the standard manner to lower the risk of graft-vs-host disease (GVHD), a reaction of the donor's immune cells against the recipient's body.

The allogeneic stem cells (bone marrow or peripheral blood stem cells) will also be given through the CVC. You will receive the drug G-CSF (filgrastim) as an injection under the skin once a day, starting 1 week after the transplant, until your blood cell levels return to normal.

Patients usually stay in the hospital for about 4 weeks after stem cell transplantation. After you are released from the hospital, you will continue to be monitored as an outpatient for infections and transplant-related complications for at least 100 days after the transplant.

You will have blood tests (about 4 tablespoons of blood) and bone marrow aspirations performed at 1, 3, 6, and 12 months after the transplant, to check if the disease is in remission (has not come back). Your health status will be followed with the help of your local doctor to find out if the leukemia or MDS comes back, as well as to check the length of your survival.

This is an investigational study. All of the drugs used in this study are approved by the FDA for treatment of cancer. Busulfan has been approved for use in stem cell transplantation. The use of these drugs together with stem cell transplant is experimental. Up to 70 patients will take part in this study. All will be enrolled at the M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis or 1) Acute myeloid leukemia past first remission, in first or subsequent relapse, or induction failures, 2) Myelodysplastic syndromes with intermediate or high risk International Prognostic Scoring System score (IPSS scores) (16), and having failed previous chemotherapy, or 3) Chronic Myeloid Leukemia, Philadelphia-chromosome positive and having failed / being resistant to therapy based on Gleevec or other tyrosine kinase inhibitors.
2. Patient has not been administered intensive systemic chemotherapeutic drugs within 21 days prior to trial enrollment (bone marrow transplant (BMT) Day -9). Gleevec, alternative tyrosine kinase inhibitors, other nonmyelosuppressive agents, low dose cytarabine, hydroxyurea is permitted if indicated to control the leukemia. All tyrosine inhibitor- or other non-myelosuppressive agents have to be terminated at least one week prior to admission for this treatment.
3. No uncontrolled infection. Protocol principal investigator (PI) will be final arbiter if there is uncertainty regarding whether a previous infection is resolved on appropriate antibiotics therapy.
4. age </= 60
5. A related or unrelated donor who is HLA-matched or mismatched in 1 HLA, A, B, C, DR or DQ locus is acceptable (i.e. at least a 9/10 matched related or unrelated donor, matched with molecular high-resolution technique per current standard for the BMT program).
6. ZUBROD performance status <2
7. Life expectancy is not severely limited by concomitant illness.
8. Left ventricular ejection fraction >/=45% No uncontrolled arrhythmias or symptomatic cardiac disease.
9. Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and carbon monoxide diffusing capacity (DLCO) >/= 50% of expected corrected for hemoglobin. In patients </= 7 years pulmonary function will be assessed per pediatric BMT routine
10. Serum creatinine </= 1.5 mg%.
11. Serum glutamic pyruvic transaminase (SGPT) </= 200 IU/ml, serum bilirubin and alkaline phosphatase within accepted laboratory standard normal limits or considered not clinically significant. No evidence of chronic active hepatitis or cirrhosis. If positive hepatitis serology, discuss with Study Chairman and perform liver biopsy pror to determining study eligibility.
12. Female patient is not pregnant (negative human chorionic gonadotropin (hCG) pregnancy test in all women of child-bearing-potential in accordance with departmental routine).
13. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.

Exclusion Criteria:

1. Effusion or ascites estimated to be >1L prior to drainage.
2. HIV-positive.
3. Hepatitis C or HBsAg positive
4. Prior stem cell transplant after a myeloablative conditioning program (such as busulfan-based using a total dose of >/= 12 mg/kg given by mouth or >/= 10 mg/kg IV, or a total-body irradiation-based program.
5. Active or prior Central Nervous System (CNS) leukemia
6. Biphenotypic acute leukemia.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2006-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Andersson BS, Valdez BC, de Lima M, Wang X, Thall PF, Worth LL, Popat U, Madden T, Hosing C, Alousi A, Rondon G, Kebriaei P, Shpall EJ, Jones RB, Champlin RE. Clofarabine +/- fludarabine with once daily i.v. busulfan as pretransplant conditioning therapy for advanced myeloid leukemia and MDS. Biol Blood Marrow Transplant. 2011 Jun;17(6):893-900. doi: 10.1016/j.bbmt.2010.09.022. Epub 2010 Oct 11. PMID 20946966
- See also: UT MD Anderson Cancer Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: September 25, 2006 to March 30, 2011. All participants were recruited at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 72 enrolled participants, one participant was not eligible and not treated. In the initial phase, the first 20 participants were fairly randomized to each of the 4 treatment arms. The rest of the participants were adaptively randomized among the arms in period 2.
Period: Initial Phase Randomization
Arm/Group | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine | Arm 4: Busulfan + Clofarabine
Started | 5 | 4 | 5 | 6
Completed | 4 | 3 | 4 | 5
Not Completed | 1 | 1 | 1 | 1
Not completed — Disease Progression | 0 | 1 | 1 | 0
Not completed — No Response | 1 | 0 | 0 | 1
Period: Adaptive Randomization
Arm/Group | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine | Arm 4: Busulfan + Clofarabine
Started | 13 | 3 | 24 | 11
Completed | 12 | 2 | 23 | 10
Not Completed | 1 | 1 | 1 | 1
Not completed — Not Evaluable | 1 | 0 | 0 | 1
Not completed — No Response | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine | Arm 4: Busulfan + Clofarabine | Total
Number analyzed (Participants) | 18 | 7 | 29 | 17 | 71
Age, Continuous [Median (Full Range); unit: years] | 33 [6 to 59] | 54 [11 to 59] | 38 [14 to 59] | 47 [7 to 59] | 46 [6 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 14 | 6 | 31
  Male | 8 | 6 | 15 | 11 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 4 | 3 | 15
  Not Hispanic or Latino | 10 | 6 | 24 | 14 | 54
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 15 | 6 | 26 | 17 | 64
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 7 | 29 | 17 | 71

OUTCOME MEASURES:

1. Primary Outcome: Treatment Related Mortality
Description: Number of participants with treatment related mortality (death) within the first 30 days following transplantation.
Time Frame: First 30 Days
Measure: Number; unit: participants
Arm/Group | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine | Arm 4: Busulfan + Clofarabine
Number analyzed (Participants) | 13 | 3 | 24 | 11
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment period defined as BMT Day -9 through BMT Day +28, post study surveillance defined as BMT Day +29 through +100. Thereafter, participant status/survival data collected quarterly as available. End of active treatment is day of stem cell infusion.
Arm/Group | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine | Arm 4: Busulfan + Clofarabine
All-Cause Mortality (participants affected / at risk) | 2/71 | 1/71 | 4/71 | 1/71
Serious Adverse Events (participants affected / at risk) | 15/71 | 6/71 | 27/71 | 15/71
Other Adverse Events (participants affected / at risk) | 18/72 | 7/72 | 29/72 | 16/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine (N=71) | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine (N=71) | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine (N=71) | Arm 4: Busulfan + Clofarabine (N=71)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
AL OTH (General disorders) | 0 | 0 | 0 | 0
ALK increased (Investigations) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0
ALT increased (Investigations) | 7 | 0 | 6 | 5
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0
AST increased (Investigations) | 0 | 0 | 0 | 0
Bacterial (Infections and infestations) | 4 | 3 | 13 | 6
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0
BOOP (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0
Broncholitis obliterans (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0
Chronic GVHD (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 1 | 1 | 0 | 0
DAH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dysrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0
Ejection fraction decreased (Cardiac disorders) | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 3 | 15 | 8
Fever (General disorders) | 0 | 0 | 2 | 0
Fluid overload (General disorders) | 0 | 0 | 2 | 0
Fungal (Infections and infestations) | 0 | 0 | 2 | 0
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
GI FIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GI OTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 | 0 | 2 | 0
HP OTH (Hepatobiliary disorders) | 0 | 0 | 0 | 0
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 2 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Low granulocyte (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Low platelet (Investigations) | 4 | 0 | 4 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NE COR (Nervous system disorders) | 0 | 0 | 0 | 0
NE PAI (Nervous system disorders) | 0 | 0 | 0 | 0
Ocular GvHD (Eye disorders) | 0 | 0 | 0 | 0
Oral GvHD (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Oral mucositis (Gastrointestinal disorders) | 1 | 0 | 6 | 1
Parasite (Infections and infestations) | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0
Peripheral neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 3
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
T bilirubin increased (Investigations) | 2 | 1 | 3 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0
Viral (Infections and infestations) | 4 | 0 | 4 | 1
VOD (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Arm 1: Busulfan + Fludarabine (30 mg/m^2) + Clofarabine (N=72) | Arm 2: Busulfan + Fludarabine (20 mg/m^2) + Clofarabine (N=72) | Arm 3: Busulfan + Fludarabine (10 mg/m^2) + Clofarabine (N=72) | Arm 4: Busulfan + Clofarabine (N=72)
Abdominal pain (Gastrointestinal disorders) | 3/71 | 3/71 | 1/71 | 1/71
AL OTH (General disorders) | 0/71 | 0/71 | 1/71 | 0/71
ALK increased (Investigations) | 3/71 | 0/71 | 5/71 | 3/71
Allergic reaction (Immune system disorders) | 0/71 | 0/71 | 2/71 | 0/71
ALT increased (Investigations) | 10/71 | 1/71 | 10/71 | 5/71
Anorexia (Metabolism and nutrition disorders) | 0/71 | 0/71 | 0/71 | 0/71
Anxiety (Psychiatric disorders) | 0/71 | 0/71 | 1/71 | 0/71
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/71 | 0/71 | 1/71 | 0/71
AST increased (Investigations) | 0/71 | 0/71 | 2/71 | 0/71
Bacterial (Infections and infestations) | 3/71 | 2/71 | 5/71 | 2/71
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 0/71 | 0/71 | 0/71 | 0/71
Blurred vision (Eye disorders) | 1/71 | 1/71 | 0/71 | 0/71
Bone pain (Musculoskeletal and connective tissue disorders) | 1/71 | 1/71 | 0/71 | 1/71
BOOP (Respiratory, thoracic and mediastinal disorders) | 0/71 | 0/71 | 0/71 | 0/71
Broncholitis obliterans (Respiratory, thoracic and mediastinal disorders) | 0/71 | 0/71 | 0/71 | 1/71
Chest pain (Cardiac disorders) | 0/71 | 1/71 | 0/71 | 0/71
Chronic GVHD (Skin and subcutaneous tissue disorders) | 1/71 | 0/71 | 0/71 | 0/71
Confusion (Psychiatric disorders) | 1/71 | 1/71 | 0/71 | 0/71
Creatinine increased (Investigations) | 2/71 | 2/71 | 0/71 | 4/71
DAH (Respiratory, thoracic and mediastinal disorders) | 0/71 | 0/71 | 0/71 | 0/71
Diarrhea (Gastrointestinal disorders) | 8/71 | 5/71 | 0/71 | 7/71
Dizziness (Nervous system disorders) | 0/71 | 0/71 | 0/71 | 0/71
Dry eye (Eye disorders) | 4/71 | 0/71 | 0/71 | 7/71
Dry skin (Skin and subcutaneous tissue disorders) | 0/71 | 0/71 | 0/71 | 0/71
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/71 | 0/71 | 0/71 | 0/71
Dysrhythmia (Cardiac disorders) | 0/71 | 0/71 | 0/71 | 1/71
Ejection fraction decreased (Cardiac disorders) | 1/71 | 0/71 | 0/71 | 0/71
Encephalopathy (Nervous system disorders) | 0/71 | 0/71 | 0/71 | 0/71
Fasciitis (Musculoskeletal and connective tissue disorders) | 0/71 | 0/71 | 0/71 | 0/71
Fatigue (General disorders) | 1/71 | 0/71 | 0/71 | 0/71
Febrile neutropenia (Blood and lymphatic system disorders) | 1/71 | 3/71 | 0/71 | 0/71
Fever (General disorders) | 7/71 | 3/71 | 12/71 | 7/71
Fluid overload (General disorders) | 2/71 | 0/71 | 0/71 | 3/71
Fungal (Infections and infestations) | 3/71 | 0/71 | 4/71 | 2/71
Gastrointestinal bleeding (Gastrointestinal disorders) | 0/71 | 0/71 | 0/71 | 0/71
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0/71 | 0/71 | 0/71 | 0/71
GI FIS (Gastrointestinal disorders) | 0/71 | 0/71 | 0/71 | 0/71
GI OTH (Gastrointestinal disorders) | 0/71 | 0/71 | 0/71 | 0/71
Hallucination (Psychiatric disorders) | 1/71 | 0/71 | 0/71 | 0/71
Headache (Nervous system disorders) | 6/71 | 2/71 | 7/71 | 5/71
Hemorrhagic Cystitis (Renal and urinary disorders) | 3/71 | 2/71 | 7/71 | 5/71
HP OTH (Hepatobiliary disorders) | 0/71 | 0/71 | 0/71 | 0/71
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 0/71 | 0/71 | 0/71 | 0/71
Hyperglycemia (Metabolism and nutrition disorders) | 1/71 | 0/71 | 1/71 | 3/71
Hypertension (Vascular disorders) | 1/71 | 2/71 | 2/71 | 0/71
Hypomagnesemia (Metabolism and nutrition disorders) | 0/71 | 0/71 | 1/71 | 0/71
Hypotension (Vascular disorders) | 0/71 | 0/71 | 0/71 | 0/71
Infusion related reaction (Injury, poisoning and procedural complications) | 1/71 | 0/71 | 0/71 | 0/71
Low granulocyte (Blood and lymphatic system disorders) | 0/71 | 0/71 | 0/71 | 0/71
Low platelet (Investigations) | 0/71 | 0/71 | 0/71 | 0/71
Myocardial infarction (Cardiac disorders) | 0/71 | 0/71 | 0/71 | 0/71
Nausea (Gastrointestinal disorders) | 18/71 | 6/71 | 27/71 | 16/71
NE COR (Nervous system disorders) | 0/71 | 0/71 | 0/71 | 0/71
NE PAI (Nervous system disorders) | 0/71 | 0/71 | 0/71 | 0/71
Ocular GvHD (Eye disorders) | 0/71 | 0/71 | 0/71 | 1/71
Oral GvHD (Gastrointestinal disorders) | 0/71 | 0/71 | 0/71 | 1/71
Oral mucositis (Gastrointestinal disorders) | 17/71 | 6/71 | 23/71 | 14/71
Parasite (Infections and infestations) | 0/71 | 0/71 | 0/71 | 0/71
Pericarditis (Cardiac disorders) | 1/71 | 0/71 | 0/71 | 0/71
Peripheral neuropathy (Nervous system disorders) | 2/71 | 1/71 | 1/71 | 0/71
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/71 | 0/71 | 4/71 | 0/71
Psychosis (Psychiatric disorders) | 0/71 | 0/71 | 4/71 | 0/71
Rash (Skin and subcutaneous tissue disorders) | 15/71 | 4/71 | 19/71 | 11/71
Skin discoloration (Skin and subcutaneous tissue disorders) | 0/71 | 0/71 | 0/71 | 1/71
Somnolence (Nervous system disorders) | 0/71 | 0/71 | 0/71 | 0/71
T bilirubin increased (Investigations) | 3/71 | 0/71 | 4/71 | 5/71
Thromboembolic event (Vascular disorders) | 0/71 | 0/71 | 1/71 | 0/71
Tinnitus (Ear and labyrinth disorders) | 1/71 | 0/71 | 0/71 | 0/71
Vaginal dryness (Reproductive system and breast disorders) | 0/71 | 0/71 | 1/71 | 1/71
Viral (Infections and infestations) | 6/71 | 3/71 | 17/71 | 6/71
VOD (Hepatobiliary disorders) | 0/71 | 0/71 | 0/71 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No